CLINICAL TRIAL: NCT00870441
Title: A Phase 1, Randomized, Double-Blind, Multiple Dose, Multi-Center Study to Compare the Safety of ASP2151 to Valacylcovir and Placebo in Healthy Male and Female Subjects
Brief Title: Study Comparing the Safety of ASP2151 to Valacyclovir and Placebo in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to treatment-emergent serious adverse events
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 15L-CL-019
Record Dates: First submitted 2009-03-25; First posted 2009-03-27 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2010-06

CONDITIONS: Safety of ASP2151
Keywords: ASP2151; Valacyclovir; Healthy Volunteers
MeSH Terms: interventions — ASP2151; Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. ASP2151 (Experimental)
  Interventions: Drug: ASP2151
- 2. Valacyclovir (Active Comparator)
  Interventions: Drug: Valacyclovir
- 3. Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP2151 — Oral
  Arms: 1. ASP2151
Drug: Valacyclovir — Oral
  Other Names: Valtrex
  Arms: 2. Valacyclovir
Drug: Placebo — Oral
  Arms: 3. Placebo

SUMMARY:
The objective of the study is to compare the safety of ASP2151 to valacyclovir and placebo in healthy male and female adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject weighing at least 45 kg with a Body Mass Index (BMI) of 18-35 kg/m2, inclusive
* If female, subject is using a medically acceptable contraceptive method along with a double-barrier method to prevent pregnancy and agrees to continue using this method throughout study; and is not lactating or pregnant as documented by a negative serum pregnancy test
* The subject is medically healthy, with a normal 12-lead electrocardiogram (ECG)

Exclusion Criteria:

* History of any clinically significant disease or malignancy excluding non-melanoma skin cancer
* History of liver disease, liver dysfunction, liver enzyme elevations, or Gilbert's disease
* History of acute or chronic pancreatitis or pancreatic insufficiency
* History of gout, hyperuricemia, or crystalluria
* History of chronic pain requiring medical therapy
* Positive test for hepatitis C virus (HCV) antibody or hepatitis B surface antigen (HBsAg)
* Positive test for human immunodeficiency virus (HIV) antibody
* Clinical laboratory tests outside the normal limits and considered by the investigator to be clinically significant
* The subject has difficulty swallowing tablets
* Clinically significant illness within one month prior to study drug administration
* History of drug or alcohol abuse within 2 years prior to study drug administration
* Treatment with prescription medication (with the exception of contraceptives and hormone replacement therapy (HRT)) or complementary and alternative medicines (CAM) within 14 days; over-the-counter products with exception of ibuprofen within 14 days; or alcohol, grapefruit or grapefruit juice containing beverage within 72 hours
* Donated blood or has had significant blood loss within 56 days prior to study drug administration or has donated plasma within 7 days prior to study drug administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Assessment of clinical laboratory evaluations and adverse events | Days 1,4,7,10,14,17,21,24, 28 and follow-up visit

SECONDARY OUTCOMES:
Assessment of ECG, vital signs and physical examination | Days 1,4,7,10,14,17,21,24 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (5):
- United States (5):
  - Daytona Beach, Florida
  - Honolulu, Hawaii
  - Evansville, Indiana
  - Austin, Texas
  - Dallas, Texas